CLINICAL TRIAL: NCT00279578
Title: Clot Formation and Clot Stability in Patients With Severe Haemophilia A - Effect of Recombinant Factor VIII and Tranexamic Acid
Brief Title: Clot Formation and Clot Stability in Patients With Severe Haemophilia A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050184
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-11-16 (Estimated); Status verified 2006-11

CONDITIONS: Hemophilia A
Keywords: haemophilia A; thrombelastography; recombinant factor VIII; thrombin generation
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII SQ; Factor VIII; Tranexamic Acid

INTERVENTIONS:
Drug: ReFacto (Recombinant factor VIII) and Tranexamic acid

SUMMARY:
In the present study we are examining the clot formation and clot stability in patients with severe haemophilia A after they receive recombinat factor VIII and after addition of tranexamic acid. Our hypothesis is that addition of tranexamic increases the clot stability. The perpective of the study is to document whether it is relevant to use traneksamic acid in surgery in patients with severe haemophilia A.

DETAILED DESCRIPTION:
In the present study we are examining the clot formation and clot stability in patients with severe haemophilia A after they receive recombinat factor VIII and after addition of tranexamic acid. Our hypothesis is that addition of tranexamic increases the clot stability. The perpective of the study is to document whether it is relevant to use traneksamic acid in surgery in patients with severe haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Severe haemophilia A
* Above 17 years old
* Thrombocyt count above 100 x 109/l within the past two years

Exclusion Criteria:

* Received recombinant factor VIII with in the past 3 days
* Inhibitor against recombinant factor VIII
* HIV-positive
* Ongoing treatment for hepatitis C
* Known kidney disease
* Allergy against Tranexamic acid
* Not able to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8
Dates: Start 2006-01; Study Completion 2006-06

PRIMARY OUTCOMES:
Clot stability

SECONDARY OUTCOMES:
clot formation,thrombine generation

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Hvas, MD, Ph.D., Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Clinical Biochemistry, Center for Haemophilia and Thrombosis, Aarhus, Denmark